CLINICAL TRIAL: NCT00118885
Title: Behavioral Intervention for Herpes Zoster Risk in Aging
Brief Title: Shingles: Immune Effects of Tai Chi
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: AG0029; R01AG018367 (NIH)
Record Dates: First submitted 2005-07-08; First posted 2005-07-12 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2006-11

CONDITIONS: Aging; Herpes Zoster
Keywords: Shingles; depression; varicella zoster virus; alternative medicine; psychoneuroimmunology
MeSH Terms: conditions — Herpes Zoster; Depression; Chickenpox

INTERVENTIONS:
Behavioral: Tai Chi Chih

SUMMARY:
The purpose of this trial is to evaluate the effects of Tai Chi Chih versus Health Education on shingles immunity in older adults as measured by unstimulated and vaccine-stimulated responses. The secondary goal of the study is to determine the effects of Tai Chi Chih versus Health Education on measures of health functioning, depressive symptoms, and health behaviors in the elderly.

DETAILED DESCRIPTION:
Shingles, also known as herpes zoster (HZ), is more common in older persons due to the weakening of the immune system with advancing age. Psychosocial stresses in the older adult also correlate with the decline in immunity. In addition, preliminary data indicate that the presence of depressive symptoms in older adults is associated with a decline in the response to varicella zoster virus (VZV) vaccination. Taken together, the untoward effects of age and depressive symptoms on VZV immunity raise the question as to whether a behavioral intervention might augment VZV specific immunity in the older adult.

Preliminary data has shown that administration of a relaxation-response based intervention, Tai Chi Chih (TCC), results in improvements in health functioning and VZV immunity in older adults as compared to a control group. TCC is a slow moving meditation comprised of twenty separate standardized movements for use in elderly populations. By standardization of training and practice schedules, TCC offers an important advantage over prior relaxation response based therapies. This controlled trial has 3 goals:

1. determine whether the practice of TCC for 16 weeks influences unstimulated- and vaccine-stimulated VZV specific immunity in adults 60 years of age and older;
2. demonstrate that TCC can produce significant changes in psychological adaptation, health behaviors, and health functioning and well-being;
3. assess whether changes in psychological adaptation, health behaviors, and health functioning correlate with changes in VZV immunity following TCC in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Older than 60 years of age at time of entry
* History of varicella or long term (>30 years) residence in the continental USA
* Accessible geographically

Exclusion Criteria:

* Immunosuppression resulting from neoplastic disease, corticosteroids or other therapy
* Significant underlying illness that would be expected to prevent completion of the study; any other condition (e.g. extensive psoriasis, chronic pain syndrome, cognitive impairment, severe hearing loss) that in the opinion of the investigator might interfere with the required evaluations
* Not ambulatory (bed-ridden)
* Prior HZ or prior receipt of varicella vaccine
* Allergic sensitivity to neomycin
* Receipt of immune globulin or other blood product within 3 months before the study period
* Receipt of other immunizations (e.g., hepatitis B vaccine) within 1 month of immunization
* Women who are not post-menopausal
* Acutely depressed or a suicidal risk
* Unable to commit to intervention schedule
* No history of varicella or varicella vaccination or no evidence of VZV immunity
* Contact with immunosuppressed individuals or pregnant women who do not have a history of chickenpox
* Active infections such as tuberculosis

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Start 2001-07; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
varicella zoster specific immunity

SECONDARY OUTCOMES:
measures of health status including SF-36 scores, depressive symptoms, and health behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Irwin, MD, Principal Investigator — Norman Cousins Professor, Cousins Center for Psychoneuroimmunology, UCLA Neuropsychiatric Institute
Locations (1):
- Cousins Center for Psychoneuroimmunology, UCLA Neuropsychiatric Institute, Los Angeles, California, United States

REFERENCES:
- [Background] Miller GE, Cohen S. Psychological interventions and the immune system: a meta-analytic review and critique. Health Psychol. 2001 Jan;20(1):47-63. doi: 10.1037//0278-6133.20.1.47. PMID 11199066
- [Background] Oxman MN, Levin MJ, Johnson GR, Schmader KE, Straus SE, Gelb LD, Arbeit RD, Simberkoff MS, Gershon AA, Davis LE, Weinberg A, Boardman KD, Williams HM, Zhang JH, Peduzzi PN, Beisel CE, Morrison VA, Guatelli JC, Brooks PA, Kauffman CA, Pachucki CT, Neuzil KM, Betts RF, Wright PF, Griffin MR, Brunell P, Soto NE, Marques AR, Keay SK, Goodman RP, Cotton DJ, Gnann JW Jr, Loutit J, Holodniy M, Keitel WA, Crawford GE, Yeh SS, Lobo Z, Toney JF, Greenberg RN, Keller PM, Harbecke R, Hayward AR, Irwin MR, Kyriakides TC, Chan CY, Chan IS, Wang WW, Annunziato PW, Silber JL; Shingles Prevention Study Group. A vaccine to prevent herpes zoster and postherpetic neuralgia in older adults. N Engl J Med. 2005 Jun 2;352(22):2271-84. doi: 10.1056/NEJMoa051016. PMID 15930418
- [Background] Irwin M, Pike J, Oxman M. Shingles Immunity and Health Functioning in the Elderly: Tai Chi Chih as a Behavioral Treatment. Evid Based Complement Alternat Med. 2004 Dec;1(3):223-232. doi: 10.1093/ecam/neh048. Epub 2004 Dec 1. PMID 15841255
- [Background] Irwin MR, Pike JL, Cole JC, Oxman MN. Effects of a behavioral intervention, Tai Chi Chih, on varicella-zoster virus specific immunity and health functioning in older adults. Psychosom Med. 2003 Sep-Oct;65(5):824-30. doi: 10.1097/01.psy.0000088591.86103.8f. PMID 14508027
- [Derived] Irwin MR, Olmstead R. Mitigating cellular inflammation in older adults: a randomized controlled trial of Tai Chi Chih. Am J Geriatr Psychiatry. 2012 Sep;20(9):764-72. doi: 10.1097/JGP.0b013e3182330fd3. PMID 21934474
- [Derived] Irwin MR, Olmstead R, Motivala SJ. Improving sleep quality in older adults with moderate sleep complaints: A randomized controlled trial of Tai Chi Chih. Sleep. 2008 Jul;31(7):1001-8. PMID 18652095